CLINICAL TRIAL: NCT05814250
Title: Is Ultrasonography Mandatory in All Children at Their First Febrile Urinary Tract Infection?
Brief Title: Ultrasonography in Children With First Febrile Urinary Tract Infection
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 01/22
Record Dates: First submitted 2023-03-28; First posted 2023-04-14 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Urinary Tract Infections
Keywords: Urinary tract infection; Kidney ultrasound; Congenital anomalies of the kidney and urinary tract
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In recent decades, different tests have been recommended by guidelines in the management of first febrile urinary tract infection (fUTI) in children, including kidney ultrasound (KUS), cystography (VCUG) and renal scintigraphy in order to exclude underlying kidney anomalies. The majority of guidelines, continue to recommend a routine KUS for all children at the first fUTI. On the other hand, as this approach is not based on robust evidence, other guidelines suggest that KUS should only be performed on selected patients according to specific risks. Despite being a non-invasive and radiation-free method, KUS tests negative in 83% of cases of fUTIs and possesses low specificity for low grade vesico-ureteral reflux (VUR). Since VUR is the most commonly associated renal malformation with UTI, it is evident that all the guidelines focus on the research of VUR, especially in times when antenatal ultrasound allows to screen for major congenital anomalies of kidney and urinary tract (CAKUT). However, VUR-associated nephropathy appears to be related to primary dysplastic damage rather than to be secondary to the reflux itself and not preventable from antibiotic prophylaxis in terms of recurrence and of kidney scar. To reduce the number of normal VCUGs performed, recent evidence regarding VUR suggests that the presence of pathogens different from E. coli and UTI recurrence may help to identify children who necessitate further investigations. A preliminary retrospective monocentric study enrolling all patients aged 2 to 36 months diagnosed with first fUTI who subsequently underwent US evaluation of the kidneys and urinary tract, found that atypical germ and recurrence of UTI exhibits a 85% sensitivity to detect pathological ultrasound. The aim of this multicentric study is to prospectively evaluate the diagnostic accuracy of the presence of atypical germ combined with the recurrence of UTI in predicting the positivity of KUS in children aged 2 months to 3 years old with first episode of fUTI

ELIGIBILITY:
Inclusion Criteria:

- Patient with first episode of fUTI that subsequently do KUS.

Exclusion Criteria:

* patients with previous episodes of UTIs
* patients on antibiotic prophylaxis
* previous finding of malformative uropathies or cystic disease
* prenatal diagnosis of CAKUT with the following parameters: Presence of oligohydramnios, alterations in renal number, location and echo structure, bladder alteration, dilations of the renal pelvis and ureters

Ages: 2 Months to 3 Years | Sex: All
Age Groups: Child
Study Population: Children aged 2 months to 3 years with the first episode of urinary tract infection
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the diagnostic accuracy of the presence of an atypical germ combined with the possible recurrence of UTI in predicting the positivity of KUS in children aged between 2 months and 3 years with first episode of fUTI | Follow up of 2 years or until the third year of age
  Sensitivity, specificity positive and negative predictive values will be evaluated. Patient will be recruited prospectively. A first sample of urine culture can be collected from urine bag, and analyzed by urine dipstick. If urine dipstick tests positive such as positivity for leukocytes and/or nitrites, a second sample will be collected with sterile methods as clan catch or bladder catheterization. Urine culture will be performed in both urine samples. In case of a UTI a subsequent follow up is recommended with an abdominal ultrasound after one month. In case of a pathological ultrasound, the subsequent diagnostic follow up it is up to the clinician, with voiding cystography or scintigraphy. During the follow up period UTI relapses will be detected.

SECONDARY OUTCOMES:
To evaluate the diagnostic accuracy of urinary culture carried out from urinary bag vs a second sample gathered from the same patient by clean catch or bladder catheterization (gold standard) | At the time of urine collection (baseline)
  Sensitivity, specificity positive and negative predictive values will be evaluated
To evaluate the concordance of the germs found in positive urinary culture carried out from urinary bag vs clean catch or bladder catheterization gathered from the same patient | At the time of urine collection (baseline)
  The concordance of the germs found with the two different samples collections will be evaluated using the Cohen's kappa coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pennesi, MD, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (3):
- Italy (3):
  - AOU Meyer IRCCS, Florence
  - IRCCS Policlinico Cà Granda, Milan
  - IRCCS materno infantile Burlo Garofolo, Trieste

IPD SHARING:
Plan to Share IPD: No